CLINICAL TRIAL: NCT00124059
Title: A Double-Blind Study of Quetiapine Fumarate (Seroquel) for the Treatment of Type A vs.Type B Alcoholics.
Brief Title: Quetiapine Fumarate (Seroquel) for the Treatment of Alcohol Dependence.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 706689
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2013-09

CONDITIONS: Alcoholism
Keywords: alcohol dependence
MeSH Terms: conditions — Alcoholism | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Type A SERO (Experimental)
  Interventions: Drug: Seroquel
- Type B SERO (Experimental)
  Interventions: Drug: Seroquel
- Type A PLA (Placebo Comparator)
  Interventions: Drug: Placebo
- Type B PLA (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Seroquel — 400mg/day quetiapine
  Arms: Type A SERO; Type B SERO
Drug: Placebo — 400mg/day placebo
  Arms: Type A PLA; Type B PLA

SUMMARY:
The purpose of this study is to determine whether seroquel is effective in the treatment of type A and type B alcohol dependence.

DETAILED DESCRIPTION:
The purpose of this study is to obtain preliminary data regarding the safety, efficacy and tolerability of quetiapine [Seroquel (SQL)] in treating Type A vs B alcohol dependent outpatients seeking treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and 18-65 years old.
2. Has a DSM-IV diagnosis of current alcohol dependence.
3. Has either Type A or Type B alcohol dependence, determined by cut-off scores for drinking amounts per day (TLFB), depression symptoms (Hamilton Depression Rating Scale--HDRS; Hamilton, 1967), and number of childhood antisocial personality symptoms. These three variables were selected based on recently published data on alcohol subtyping by Pettinati et al., 2000b).
4. Meets the following drinking criteria, measured by TLFB: a. drink within 30 days of starting pharmacotherapy treatment, b. reports a minimum of 48 standard alcoholic drinks (avg 12 drinks/wk) in a consecutive 30-day period over the 90-day period prior to starting pharmacotherapy (i.e., a minimum of 40% days drinking), and c. has 2 or more days of heavy drinking (defined as 5 or more drinks per day in males and 4 or more drinks per day in females) in this same pre-treatment period. [Note: To be a subject in the study, the patient must have been drinking enough in the 90 days before the trial so that a baseline exists in order to then measure reductions in drinking during the trial.]
5. Prior to starting pharmacotherapy, scores below 8 on the Clinical Institutes Withdrawal Assessment for Alcohol (CIWA; Shaw et al, 1981), and has at least 3 consecutive days of abstinence, as determined by subject report, breathalyzer measures, and a collateral report.
6. Speaks, understands and prints in English.
7. Gives written informed consent.

Exclusion Criteria:

1. Has evidence of dependence on a substance other than alcohol (except nicotine), test positive on the urine drug screen (with the exception of THC) in the screening week (only one repeat testing permitted), or require inpatient detoxification for any substance.
2. Has hepatocellular disease indicated by elevations of SGPT (ALT) and SGOT (AST) of at least 4.5 times normal after the required 3 days of abstinence, or elevated bilirubin (>1.3).
3. Patients with hepatocellular disease as evidenced by AST or ALT levels at least 2 times normal who test positive on a screening test for hepatitis A, B or C.
4. Meets diagnostic criteria for a current unstable or serious psychiatric or medical illness. For example, bipolar affective disorder, schizophrenia or any other psychotic disorder, or organic mental disorder; has serious heart, lung, kidney, immune system, GI tract (ulcerative colitis, regional enteritis, or gastrointestinal bleeding) disease.
5. Has taken any psychotropic medications (or disulfiram) regularly within the last 2 weeks or needs immediate treatment with a psychotropic medication (with the exception of detoxification medications or benadryl used sparingly for sleep);
6. Tests positive on a pregnancy test, is contemplating pregnancy in the next 12 months, is nursing, or is not using an effective contraceptive method if the S is of child-bearing potential.
7. Has known hypersensitivity to antipsychotics.
8. Has participated in any investigational drug trial within 30 days prior to the study.
9. History of seizures including alcohol withdrawal seizures.
10. History of head trauma.
11. Family history of seizures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2003-03; Primary Completion 2005-09 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
TLFB (TimeLine FollowBack) for 1) proportion of days abstinent; 2) proportion of days of heavy drinking; 3) time to the return of heavy drinking (drinking heavily for 2 out of 30 days). | 13 weeks

SECONDARY OUTCOMES:
1. Patient acceptability of the pharmacotherapy (measured by treatment drop outs and pill noncompliance) 2. Changes in craving for alcohol over the course of treatment 3. Changes in any mood and anxiety symptoms over the course of treatment | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helen M Pettinati, PhD, Principal Investigator — University of Pennsylvania Treatment Research Center
Locations (1):
- University of Pennsylvania Treatment Research Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Kampman KM, Pettinati HM, Lynch KG, Whittingham T, Macfadden W, Dackis C, Tirado C, Oslin DW, Sparkman T, O'Brien CP. A double-blind, placebo-controlled pilot trial of quetiapine for the treatment of Type A and Type B alcoholism. J Clin Psychopharmacol. 2007 Aug;27(4):344-51. doi: 10.1097/JCP.0b013e3180ca86e5. PMID 17632217